CLINICAL TRIAL: NCT03345199
Title: Effects of Inspiratory Muscle Training in Persons With Advanced Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Min-Hui Huang, Associate Professor of Physical Therapy, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PP-1703-27264
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis, Inspiratory Muscle Training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory Muscle Trainer (IMT) (Experimental): Inspiratory Muscle Trainer (IMT) provides resistance as a person inhales, thereby strengthening respiratory muscles.
  Interventions: Other: Inspiratory Muscle Trainer (IMT)

INTERVENTIONS:
Other: Inspiratory Muscle Trainer (IMT) — During the 10-week training period, participants will perform exercises using a Threshold Inspiratory Muscle Trainer (IMT) at 3 sets of 15 repetitions per day. The initial resistance of the IMT unit will be at 30% of participants' maximum inspiratory pressure (MIP). Resistance for the IMT unit will be increased progressively and adjusted weekly by a licensed physical therapist based on participant's MIP at baseline, Borg perceived rate of exertion, and symptoms.

SUMMARY:
This study evaluates the effects of a 10-week inspiratory muscle training on the outcomes of respiratory muscle strength, fatigue, activity participation, and respiratory infection rates in persons with advanced Multiple Sclerosis (MS). Participants will perform daily exercise using the Threshold Inspiratory Muscle Trainer (IMT) device during the training period. The study will assess whether the participants improve after the training, and whether the effects can be maintained after the training ends.

DETAILED DESCRIPTION:
People with advanced multiple sclerosis (MS) often experience impairments in strength and endurance in the muscles of respiration. This can cause increased difficulty with breathing which may lead to increased respiratory infection. People with weak respiratory muscles may need to use more effort for breathing and this can be tiring and limiting a person's ability to participate in activities. Complications from breathing problems, such as pneumonia, are the most frequent reason for critical illness and intensive care in people with MS, particularly as the disease progresses.

Exercises of the respiratory muscles have the potential to improve breathing in people with MS. The goal of this study is to examine the effects of a 10-week respiratory muscle exercise program on respiratory muscle strength, fatigue, activity level, and respiratory infection rates in people with advanced MS. The study will assess whether the participants improve after the training, and whether the effects can be maintained after the training ends.

The study will invite 40 people with advanced MS to participate in a 10-week exercise program to strengthen respiratory muscles. Participants will use a device that is easy to use and provides a resistance while inhaling. Participants will perform the exercises after they receive the instruction from researchers. The progression of exercises will be tailored to each individual's tolerance to the exercise. The study will measure participants' respiratory muscle strength, perceived fatigue, participation in daily recreational activities such as coffee time, and respiratory infection rates to evaluate the effects of the program. The measurements will be done upon enrollment into the study at the baseline, after 10-week no training baseline period before the intervention, mid-point during the 10-week training, at the completion of the 10-week training, at 4 weeks and at 8 weeks after the training ends. The study will evaluate if participants improve after the training, and if the improvements can be maintained for up to 8 weeks after the training.

Outcomes from this research will help to better understand effective treatments for breathing problems in people with advanced MS. The study will be able to inform clinicians and researchers about effective protocols for respiratory muscle training in advanced MS. These results will contribute to long-term research goals, including reducing complications from respiratory problems, delaying disability associated with MS, and improving function and quality of life in people with advanced MS.

ELIGIBILITY:
Inclusion Criteria:

* Residents of The Boston Home
* Diagnosis of multiple sclerosis by a physician
* Expanded Disability Status Scale >6.5
* Able to follow instructions in English

Exclusion Criteria:

* Hospitalization for exacerbation of MS within the previous 2 months
* Unstable heart, lung, or other physical conditions
* Current smoker
* Oral temperature greater than 100 degrees Fahrenheit
* Acute illness, such as infection, inflammation, ongoing chest pain, or short of breath with light activities
* Current neurological diseases other than MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Maximal inspiratory Pressure (MIP) | Baseline to 28 weeks
  MIP will be obtained using Micro Respiratory Pressure Meter (MicroRPM). Participants will perform three trials and the best value of the three attempts will be used.
Change in Maximal Expiratory Pressure (MEP) | Baseline to 28 weeks
  MEP will be obtained using Micro Respiratory Pressure Meter (MicroRPM). Participants will perform three trials and the best value of the three attempts will be used.

SECONDARY OUTCOMES:
Change in Fatigue | Baseline to 28 weeks
  Fatigue will be measured by Modified Fatigue Impact Scale, where 0 is no impact and 20 is most severe impact on daily life
Change in Activity Participation | Baseline to 28 weeks
  The average number of recreational programs attended by each participant per day.
Change in Respiratory Infection Incidents | Baseline to 28 weeks
  The total number of incidence of respiratory infection of each participant. All incidence of respiratory infection will be documented by nursing staff.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hui Huang, PhD, Principal Investigator — University of Michigan-Flint
Locations (2):
- United States (2):
  - The Boston Home, Boston, Massachusetts
  - University of Michigan-Flint, Flint, Michigan

IPD SHARING:
Plan to Share IPD: Undecided